CLINICAL TRIAL: NCT06359613
Title: Development and Efficacy Assessment of Aglutenic Product to Improve the Nutritional Status of Celiac Children
Brief Title: Efficacy Assessment of Gluten Free Cupcakes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Veterinary and Animal Sciences, Lahore - Pakistan (Other)
Responsible Party: Principal Investigator, Shaista Jabeen, Principal Investigator, University of Veterinary and Animal Sciences, Lahore - Pakistan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 029/IRC/BMR
Record Dates: First submitted 2024-03-29; First posted 2024-04-11 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Celiac Disease in Children
Keywords: gluten sensitivity children nutritional status food choices
MeSH Terms: interventions — Food

STUDY DESIGN:
Intervention Model Description: The product will be provided to intervention group (n=50) in polyethylene bags containing 28 cupcakes (35gm by weight/cupcake, 2/day) providing approximately 20%DV of energy. Cupcakes of equal weight and size made with rice flour (mostly used recipe) will be provided to the control group (n=50)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gluten Free cupcake Group (Experimental): Nutrient rich food product (cupcakes) from flour blends of Sorghum, chickpea, Flaxseed and Almond will be prepared and flour concentration will be so adjusted to provide >20% daily value of nutrients for children of 3-8 years of age. 2 cupcakes/ day, 35g each will be provided to participants for 12 weeks.
  Interventions: Dietary Supplement: nutrient rich food product
- Placebo group (Placebo Comparator): Cupcakes from usually used gluten free rice flour will be prepared. 2 cupcakes/ day, 35g each will be provided to participants for 12 weeks.
  Interventions: Dietary Supplement: food product

INTERVENTIONS:
Dietary Supplement: nutrient rich food product — Cupcakes from flour blends of Sorghum, chickpea, Flaxseed and Almond will be prepared and flour concentration will be so adjusted to provide >20% daily value of nutrients for children of 3-8 years of age. 2 cupcakes/ day, 35g each will be provided to participants for 12 weeks.
  Arms: Gluten Free cupcake Group
Dietary Supplement: food product — Cupcakes from usually used gluten free rice flour will be prepared. 2 cupcakes/ day, 35g each will be provided to participants for 12 weeks.
  Arms: Placebo group

SUMMARY:
Randomized controlled trial will be conducted after getting informed consent form from each study participant meeting inclusion criteria (n=70, 35 control group +35 intervention group, 3-8years of age). After consumer acceptance against various attributes of aglutenic cupcake, the product will be provided in polyethylene bags containing 28 cupcakes (35gm by weight/cupcake, 2 cupcakes for each day) providing approximately 20% daily value (DV) of energy. Cupcakes of equal weight and size made with rice flour (mostly used recipe) will be provided to the control group. Further product will be provided on follow-up visits. The compliance to a gluten free diet GFD and supplemented product will be confirmed by a Food Frequency Questionnaire (FFQ).

DETAILED DESCRIPTION:
Raw Material/ Preparation of flour blends for aglutenic (gluten free) cupcakes:

Sorghum, chickpea, Flaxseed and Almond rich in healthy nutrients will be purchased from the local market. All these ingredients was ground into fine powder using uncontaminated grinder. Different flour blends was prepared by substituting whole wheat flour with Sorghum, Chickpea, Flaxseed and Almond flour at different replacement levels.

The efficacy study protocol was approved by the Bioethics Committee for randomized controlled trial (RCT). Written informed consent was obtained by the parents of children or their legal guardian.

Target population: Celiac Disease/gluten sensitive patients (n= 70, 35 control + 35 intervention) was recruited according to European Society for Pediatric Gastroenterology Hepatology and Nutrition (ESPGHAN) criteria.

Inclusion criteria:

In accordance with the inclusion criteria, boys and girls suffering from celiac disease was recruited:

* Positive trans-glutaminase antibody (tTG) as currently recommended test is the serum Immunoglobulin A (IgA) tissue trans-glutaminase antibody (tTG). The test has a sensitivity and specificity of greater than 90%.
* Clinical response to gluten free diet
* In the age range of 3-8 years

Exclusion Criteria:

* Patients on any other designed diet
* Taking vitamins and mineral supplements
* Individuals presenting with any other intestinal inflammatory disease, malignant diseases, chronic infections, thyroid, renal or hepatic alterations
* Taking drugs known to effect lipid and /or carbohydrate metabolism will be excluded from the study.

Effect of interventional product on nutritional status of participants will be assessed through anthropometric measurements, gastrointestinal complaints and following hematological indices;

* Complete Blood Count (CBC) WBCs, RBCs, MCV, Hb. , Hct. , Platelets
* Total Protein
* Lipid Profile HDL, LDL, VLDL, Cholesterol
* SGPT, SGOT
* Serum Electrolytes (Na ,Ca, K)

ELIGIBILITY:
Inclusion Criteria:

* Positive tissue trans-glutaminase antibody (tTG)
* Clinical response to gluten free diet

Exclusion Criteria:

* Vitamins and mineral supplements
* Intestinal inflammatory diseases
* Malignant diseases of intestines
* Chronic infections,
* Thyroid, renal or hepatic alterations
* Celiac patients with diabetes
* Taking drugs known to effect lipid and /or carbohydrate metabolism

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2020-01-03 (Actual)

PRIMARY OUTCOMES:
Body Weight | 12 weeks
  Body weight (in kilograms) will be measured using a weight machine with standardization done after every 20 readings.
Height of the patients | 12 weeks
  Height (in centimeters) will be measured (without shoes) in the position, back and hips touching the wall by using wall mounted stedio-meter
Mid upper Arm Circumference (MUAC) | 12 weeks
  Mid-upper arm circumference (MUAC) in centimeters will be measured midpoint between the acromion process of the scapula and the tip of the elbow.
Body Mass Index (BMI) | 12 weeks
  BMI will be calculated by using standard formula as weight in kilograms divided by height in meter square kg/m2. World Health Organization (WHO) standard growth charts, designed separately for boys and girls will be used as a research tool to assess the nutritional status.
Complete Blood Count (CBC) | 12 weeks
  White Blood Cells 10^9/L Red Blood Cells million/mm3 Mean Corpuscular Volume 10^6/µL Hemoglobin g/dL Hematocrit % Platelets 10^9/L
Total Protein | 12 weeks
  Serum Total Protein g/dL
Lipid Profile | 12 weeks
  High Density Lipoproteins mg/dL Low Density Lipoproteins mg/dL Very Low-Density Lipoproteins mg/dL Serum Total Cholesterol mg/dL
Liver Enzymes | 12 weeks
  serum glutamic-pyruvic transaminase SGPT- U/L, serum glutamic-oxaloacetic transaminase SGOT-U/L
Serum Electrolytes | 12 weeks
  Sodium mmol/L Calcium mg/dL Potassium mmol/L

SECONDARY OUTCOMES:
Gastrointestinal Symptoms | 12 weeks
  Rate of diarrhea, constipation, Severity of abdominal pain, steatorrhea, flatulence and appetite will be monitored by using Gastrointestinal Rating Scale with addition of Steatorrhea.

CONTACTS AND LOCATIONS:
Overall Officials: Shaista Jabeen, Principal Investigator — University of Veterinay and Animal Sciences,Lahore,Pakistan
Locations (1):
- UVAS, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
study outcomes will be shared with other researchers through publication without personal identification

REFERENCES:
- [Background] Suliburska J, Krejpcio Z, Regula J, Grochowicz A. Evaluation of the content and the potential bioavailability of minerals from gluten-free products. Acta Sci Pol Technol Aliment. 2013 Jan-Mar;12(1):75-9. PMID 24584867